CLINICAL TRIAL: NCT01401985
Title: A Single-Blind, Pilot Study to Determine the Tolerability and Safety of TD-1211 in Subjects With Opioid-Induced Constipation
Brief Title: A Study of TD-1211 in Subjects With Opioid-Induced Constipation (OIC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TD-1211-0076
Record Dates: First submitted 2011-07-19; First posted 2011-07-26 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Opioid Induced Constipation
Keywords: Opioid induced constipation; OIC; Constipation; Opioid side effects; morphine induced constipation
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — 3-(8-(2-(cyclohexylmethyl(2,3-dihydroxypropionyl)amino)ethyl)-8-azabicyclo(3.2.1)oct-3-yl)benzamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): 5 mg TD-1211 once daily for 4 days followed by 10 mg for 14 days
  Interventions: Drug: TD-1211
- Cohort 2 (Experimental): 5 mg TD-1211 once daily for 4 days followed by 15 mg for 14 days
  Interventions: Drug: TD-1211
- Cohort 3 (Experimental): 5 mg TD-1211 once daily for 2 days followed by 10 mg for 14 days
  Interventions: Drug: TD-1211
- Cohort 4 (Experimental): 5 mg TD-1211 once daily for 2 days followed by 15 mg for 14 days
  Interventions: Drug: TD-1211
- Cohort 5 (Experimental): 2 mg TD-1211 once daily for 14 days
  Interventions: Drug: TD-1211; Drug: Placebo
- Cohort 6 (Experimental): 2.5 mg TD-1211 every 6 hours for 14 days
  Interventions: Drug: TD-1211; Drug: Placebo

INTERVENTIONS:
Drug: TD-1211 — Capsules
Drug: Placebo — Capsules
  Arms: Cohort 5; Cohort 6

SUMMARY:
A Single-Blind, Pilot Study to Determine the Tolerability and Safety of TD-1211 in Subjects with Opioid-Induced Constipation

ELIGIBILITY:
Inclusion Criteria:

* stable dose of opioids for at least 12 weeks before screening visit
* less than or equal to 5 spontaneous bowel movements for a 2 week period and experiencing at least one other symptom of constipation
* willing to stop laxatives and other bowel treatments; rescue laxative allowed

Exclusion Criteria:

* Clinically significant condition or illness (other than the condition for which the pain medication was prescribed)
* Have participated in another clinical trial of an investigational drug 30 days prior to screening
* History of cancer treatment except adequately treated localized skin cancer within 5 years of screening
* History of chronic constipation prior to opioid therapy
* Females who are pregnant or breast feeding
* Have any condition that may affect drug absorption (e.g. previous GI surgery)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TD-1211 | 14 days

SECONDARY OUTCOMES:
Complete spontaneous bowel movements (CSBM); Spontaneous bowel movements (SBM) | Weekly assessments throughout Treatment Period
  Change from baseline in the weekly SBM and CSBM frequency

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Theravance Biopharma Investigational Site, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.